CLINICAL TRIAL: NCT03362463
Title: Long-Term Follow-Up and Management Patterns of Patients With Acute Coronary Syndrome in Middle East and Africa
Acronym: TOURACO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00256
Record Dates: First submitted 2017-11-06; First posted 2017-12-05 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Acute Coronary Syndrom

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Acute Coronary Syndrom: acute coronary syndrome in a real-life setting for patients hospitalized with an ACS (i.e. STEMI, NSTEMI, unstable angina)
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
A multinational, prospective and observational study that will assess the management of ACS in real-life practices in Middle East North Africa area.

DETAILED DESCRIPTION:
The aim of this Middle Eastern and African study is to describe the short- and long-term (i.e. up to 3 years following the index event) management in patients hospitalized for an Acute Coronary Syndrome and pharmacological management patterns in a 'real-life' setting.

The TOURACO observational study will include not only hospitals with cardiac intervention facilities but also regional and community-type hospitals that have limited (if at all) cardiac intervention facilities. The treatments prescription will be left to the investigator discretion, and will be used in accordance with the local label of each country. Off-label medication is not authorized in TOURACO study.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting to the emergency room (or equivalent) and diagnosed with UA, STEMI or NSTEMI will be eligible to participate if all the following criteria apply:

1. Provision of subject informed consent.
2. Contact Order Form has been provided.
3. Female and/or male aged 18 years and over.
4. Diagnosis of STEMI, NSTEMI or UA using the following definitions:

   Criteria for STEMI diagnosis :
   1. History of chest pain/discomfort, and
   2. Persistent ST-segment elevation (> 30 min) of ≥ 0.1 mV in 2 or more contiguous ECG leads or presumed new left bundle branch block (LBBB) on admission, and
   3. Elevation of cardiac biomarkers (CK-MB, troponins): at least one value above the 99th percentile of the upper reference limit.

   Criteria for NSTEMI diagnosis :

   (a) History of chest pain/discomfort, and (d) Lack of persistent ST-segment elevation, LBBB or intraventricular conduction disturbances, and (e) Elevation of cardiac biomarkers (CK-MB, troponins): at least one value above the 99th percentile of the upper reference limit.

   Criteria for Unstable Angina diagnosis :
   1. Symptoms of angina at rest or on minimal exercise, and
   2. (Transient) ST-T changes, and
   3. No significant increase in biomarkers of necrosis but objective evidence of ischemia by non-invasive imaging or significant coronary stenosis (at angiography).
5. Hospitalized within 24 hours of onset of symptoms during the current episode* or transferred from another hospital within 24 hours of the onset of symptoms**.

   * In case of intermittent symptoms, the symptoms onset is that of the last episode ** If the referred hospital can get the initial data of the patient from the transferring hospital, transferring period is not considered as a limitation for patient initiation

Exclusion Criteria:

Patients will not be eligible to participate if any of the following exclusion criteria are present:

1. UA, STEMI and NSTEMI precipitated by or as a complication of surgery, trauma, or gastrointestinal bleeding or post-PCI.
2. UA, STEMI and NSTEMI occurring in patients already hospitalized for other reasons.
3. Presence of any condition/circumstance which in the opinion of the Investigator could significantly limit the complete follow-up of the patient (i.e. tourist, nonnative speaker or does not understand the local language, psychiatric disturbances).
4. Already included in TOURACO observational study by another center/investigator.
5. Presence of serious/severe co-morbidities in the opinion of the Investigator which may limit short-term (i.e. 6 months) life expectancy.
6. If participating in any interventional clinical trial, should be adapted to each country local regulation.
7. Patients with any psychotic disorders.
8. Pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the emergency room (or equivalent) and diagnosed with UA, STEMI or NSTEMI.
Sampling Method: Non-Probability Sample
Enrollment: 1191 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Antithrombotic includinhg Dual Antiplatelet(DAPT) Treatment patterns | 1 Month
  Prescription of Antithrombotic including Dual Antiplatelet(DAPT) Treatment patterns at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)
Antihypertensive as apart of ACS Treatment patterns | 1 Month
  Prescription of Antihypertensive as apart of ACS Treatment patterns at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)
Diabetic lowering agents as a part of ACS Treatment patterns in the ACS patients with Diabetes including Type 2 DM | 1 Month
  Prescription of Diabetic lowering agents as a part of ACS Treatment patterns in the ACS patients with Diabetes including Type 2 DM at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)
Cholesterol lowering agents including statins as a part of ACS Treatment patterns | 1 Month
  Prescription of cholesterol lowering agents including statins as a part of ACS Treatment patterns at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)

SECONDARY OUTCOMES:
Antithrombotic includinhg Dual Antiplatelet(DAPT) Treatment patterns | 6 Month
  Prescription of Antithrombotic including Dual Antiplatelet(DAPT) Treatment patterns at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)
level of control of the different ACS related risk factor | 1,6,12,24 & 36 Month
  Level of control of ACS risk factors (diabetes, HT and dyslipidemia) at intrahospital period (from the first contact till discharge), and at 6 months of follow up. At 12, 24 and 36 months, the level will be measured if the patient comes for a planned visit.
Deviation of the treatment patterns of ACS | 3 Years
  Deviation of the treatment patterns of ACS against what is recommended in the local guidelines for the management of ACS at the different time intervals
Antihypertensive as apart of ACS Treatment patterns | 6,12,24 & 36 Months
  Prescription of Antihypertensive as apart of ACS Treatment patterns at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)
Antithrombotic includinhg Dual Antiplatelet(DAPT) Treatment patterns | 1 Year
  Prescription of Antithrombotic including Dual Antiplatelet(DAPT) Treatment patterns at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)
Antithrombotic includinhg Dual Antiplatelet(DAPT) Treatment patterns | 24 Month
  Prescription of Antithrombotic including Dual Antiplatelet(DAPT) Treatment patterns at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)
Antithrombotic includinhg Dual Antiplatelet(DAPT) Treatment patterns | 36 Month
  Prescription of Antithrombotic including Dual Antiplatelet(DAPT) Treatment patterns at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)
Diabetic lowering agents as a part of ACS Treatment patterns in the ACS patients with Diabetes including Type 2 DM | 6,12,24 & 36 Months
  Prescription of Diabetic lowering agents as a part of ACS Treatment patterns in the ACS patients with Diabetes including Type 2 DM at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)
Cholesterol lowering agents including statins as a part of ACS Treatment patterns | 6,12,24 & 36 Months
  Prescription of cholesterol lowering agents including statins as a part of ACS Treatment patterns at one month of follow-up after discharge from hospital, then confirm whether it is against international guidelines (ESC or ACC guidelines or against local guidelines when the international one are not applicable)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00256&attachmentIdentifier=a1791389-7ffc-4ac2-b519-0c5922e16e55&fileName=redacted_CSR_synopsis.pdf&versionIdentifier=